CLINICAL TRIAL: NCT01802073
Title: Treatment of Primary Sclerosing Cholangitis in Inflammatory Bowel Disease Patients With Oral Vancomycin by the Study of Its Antimicrobial and Immunomodulating Effects
Brief Title: Primary Sclerosing Cholangitis With Oral Vancomycin by the Study of Its Antimicrobial and Immunomodulating Effects
Acronym: PSC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kenneth L. Cox, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22591
Record Dates: First submitted 2013-02-21; First posted 2013-03-01 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Inflammation of the bile ducts; biliary scarring; obstruction
MeSH Terms: conditions — Cholangitis, Sclerosing; Bites and Stings | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Vancomycin (Experimental): 1) For children who weight < or = 30 kg, the vancomycin dose will be 50 mg/kg/day given orally 3 times per day for the 1st month and continue with the same dose for subsequent months if the clinical laboratory studies improved and are normal. If the laboratory studies are not normal the dose will be increased to 75 mg/kg/day given orally 3 times per day for the 2nd month and 100mg/kg/day given orally 3 times per day the 3rd month. If the laboratory studies do not improve by the end of the 3rd month since starting the vancomycin, the vancomycin will be stopped and the child will not continue the study. 2) For adults and children who weigh >30 kg, the vancomycin dose will be 500 mg given orally 3 times per day for the 1st month and continue with this dose if the clinical laboratory studies improve and are normal. If the laboratory studies are not normal the dose will be increased to 750 mg 3 times per day for the 2nd month and 1000 mg 3 times per day the 3rd month.
  Interventions: Drug: Oral Vancomycin

INTERVENTIONS:
Drug: Oral Vancomycin
  Other Names: Vancocin

SUMMARY:
Determine the benefit of oral vancomycin therapy for Primary Sclerosing Cholangitis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate changes in the fecal and salivary/urinary microbiota during vancomycin treatment of children and adults with Primary Sclerosing Cholangitis (PSC), identify features of the host microbiota that are associated with disease activity and/or response to treatment and further delineate the immunological effects of oral vancomycin treatment of PSC. This study will correlate changes in microbiota with the immunological effects of oral vancomycin in children and adults with PSC. The results of this proposal will lead to new and validated targets for diagnosis and treatment of PSC that will have high impact in the short and long term for patients and their families.

Interim results were published in Abarbanel et al, J Clin Immunol 2013 (see References).

ELIGIBILITY:
Inclusion Criteria:

* PSC Diagnosis: Liver biopsy and/or imaging (MRCP, ERCP, CT, or US
* Colonoscopy within 1 year or starting of study
* 2 groups:

  1. IBD (Inflammatory bowel disease) and PSC: details of extent and type of IBD
  2. No IBD and PSC, but positive p-ANCA or ASCA serologies indicating possible IBD.

Exclusion Criteria:

* Allergy to Vancomycin
* PSC not associated with IBD or NO positive IBD antibodies (p-ANCA [anti- neutrophil cytoplasmic antibody] or ASCA [anti-Saccharomyces cerevisiae antibody])
* Cholangiocarcinoma
* On oral or topical (enemas or suppositories) corticosteroids,topical mesalamine, or biologics (infliximab, adalimumab, certolizumab).

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cox, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

REFERENCES:
- [Result] Abarbanel DN, Seki SM, Davies Y, Marlen N, Benavides JA, Cox K, Nadeau KC, Cox KL. Immunomodulatory effect of vancomycin on Treg in pediatric inflammatory bowel disease and primary sclerosing cholangitis. J Clin Immunol. 2013 Feb;33(2):397-406. doi: 10.1007/s10875-012-9801-1. Epub 2012 Oct 9. PMID 23054338
- [Derived] Ali AH, Damman J, Shah SB, Davies Y, Hurwitz M, Stephen M, Lemos LM, Carey EJ, Lindor KD, Buness CW, Alrabadi L, Berquist WE, Cox KL. Open-label prospective therapeutic clinical trials: oral vancomycin in children and adults with primary sclerosing cholangitis. Scand J Gastroenterol. 2020 Aug;55(8):941-950. doi: 10.1080/00365521.2020.1787501. Epub 2020 Jul 7. PMID 32633158
- See also: Stanford Clinical Trials — http://med.stanford.edu/clinicaltrials/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants in the adult cohort completed the study but were not analyzed for outcomes (1 post-liver transplant patient; 1 completed the study but followed a diet that could influence results analysis). Two adult participants who consented but withdrew prior to treatment were not analyzed for outcomes.
Groups:
- Oral Vancomycin-Children: For children who weight < or = 30 kg, the vancomycin dose will be 50 mg/kg/day given orally 3 times per day for the 1st month and continue with the same dose for subsequent months if the clinical laboratory studies improved and are normal. If the laboratory studies are not normal the dose will be increased to 75 mg/kg/day given orally 3 times per day for the 2nd month and 100mg/kg/day given orally 3 times per day the 3rd month. If the laboratory studies do not improve by the end of the 3rd month since starting the vancomycin, the vancomycin will be stopped and the child will not continue the study.
  Oral Vancomycin
- Oral Vancomycin-Adults: For adults and children who weigh >30 kg, the vancomycin dose will be 500 mg given orally 3 times per day for the 1st month and continue with this dose if the clinical laboratory studies improve and are normal. If the laboratory studies are not normal the dose will be increased to 750 mg 3 times per day for the 2nd month and 1000 mg 3 times per day the 3rd month.
  Oral Vancomycin
Period: Overall Study
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
Started | 14 | 20
Completed | 9 | 9
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliant | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 7

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Customized [Count of Participants; unit: Participants]
  0-6 years | 2 | 0 | 2
  7-12 years | 5 | 0 | 5
  13-17 years | 6 | 0 | 6
  18-64 years | 1 | 20 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 8 | 18 | 26

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Elevated Alanine Aminotransferase (ALT) at Baseline and With Clinically Significant Improvement at Month 3
Description: Clinically significant improvement was determined by investigator assessment per participant based on their medical history and disease stage. Elevated ALT was any value greater than the upper limit of the standard reference range used by patient's laboratory.
Time Frame: Baseline; Month 3
Population: Participants with ALT elevated at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
Number analyzed (Participants) | 10 | 9
Participants | 10 | 6

2. Primary Outcome: Count of Participants With Elevated Gamma-glutamyltransferase (GGT) at Baseline and With Clinically Significant Improvement at Month 3
Description: Clinically significant improvement was determined by investigator assessment per participant based on their medical history and disease stage. Elevated GGT was any value greater than the upper limit of the standard reference range used by patient's laboratory.
Time Frame: Baseline; Month 3
Population: Participants with GGT elevated at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
Number analyzed (Participants) | 8 | 9
Participants | 8 | 6

3. Primary Outcome: Count of Participants With Elevated ALT and/or GGT at Baseline and With Clinically Significant Improvement at Month 3
Description: Clinically significant improvement was determined by investigator assessment per participant based on their medical history and disease stage. Elevated ALT (and GGT) was any value greater than the upper limit of the standard reference range used by patient's laboratory.
Time Frame: Baseline; Month 3
Population: Participants with ALT and/or GGT elevated at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
Number analyzed (Participants) | 10 | 10
Participants | 10 | 8

4. Primary Outcome: Count of Participants With Abnormal Magnetic Resonance Cholangiopancreatography (MRCP) Imaging at Baseline and With Clinically Significant Improvement at Year 1
Description: Clinically significant improvement was determined by investigator assessment per participant based on their medical history and disease stage. MRCP imaging was abnormal if it included biliary beading, biliary strictures, dilated bile duct, and/or liver fibrosis.
Time Frame: Baseline; Year 1
Population: Participants with abnormal MRCP at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
Number analyzed (Participants) | 8 | 8
Participants | 6 | 4

5. Primary Outcome: Count of Participants With Abnormal Liver Biopsies at Baseline and With Clinically Significant Improvement at Year 1
Description: Clinically significant improvement was determined by investigator assessment per participant based on their medical history and disease stage. Liver pathology was considered abnormal if the biopsy was S1 or greater on the liver fibrosis staging scale (S0 no fibrosis, S1 mild fibrosis, S2 moderate fibrosis, S3 sever fibrosis, S4 cirrhosis).
Time Frame: Baseline; Year 1
Population: Participants with abnormal liver biopsy at baseline and who had a post-treatment liver biopsy are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
Number analyzed (Participants) | 3 | 0
Participants | 3 | 0

6. Primary Outcome: Count of Participants With Abnormal MRCP and/or Liver Biopsy at Baseline and With Clinically Significant Improvement at Year 1
Description: Clinically significant improvement was determined by investigator assessment per participant based on their medical history and disease stage. MRCP imaging was abnormal if it included biliary beading, biliary strictures, dilated bile duct, and/or liver fibrosis. Liver pathology was considered abnormal if the biopsy was S1 or greater on the liver fibrosis staging scale (S0 no fibrosis, S1 mild fibrosis, S2 moderate fibrosis, S3 sever fibrosis, S4 cirrhosis).
Time Frame: Baseline; Year 1
Population: Participants with abnormal MRCP and/or liver biopsy at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
Number analyzed (Participants) | 10 | 9
Participants | 10 | 4

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Oral Vancomycin-Children | Oral Vancomycin-Adults
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/20
Other Adverse Events (participants affected / at risk) | 0/14 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Vancomycin-Children (N=14) | Oral Vancomycin-Adults (N=20)
Biliary stricture requiring stent (Hepatobiliary disorders) | 1 | 0
Progression of PSC (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes